CLINICAL TRIAL: NCT00697125
Title: Study to Evaluate the Immunogenicity and Reactogenicity of Various Formulations of GSK Biologicals' (Previously SmithKline Beecham Biologicals') Recombinant Hepatitis B Vaccine With Different Adjuvants in Healthy Adult Volunteers
Brief Title: Immunogenicity & Reactogenicity of Various Formulations of Recombinant Hepatitis B Vaccine With Different Adjuvants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Isabelle Harpigny, GSK
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 208129/005
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2008-06-13 (Estimated); Status verified 2008-06

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Engerix™-B; Recombinant hepatitis B vaccine
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Group A (Active Comparator)
  Interventions: Biological: Engerix™-B
- Group B (Experimental)
  Interventions: Biological: Hepatitis B vaccine, experimental formulation
- Group C (Experimental)
  Interventions: Biological: HBV-MPL vaccine (208129)

INTERVENTIONS:
Biological: Engerix™-B — Intramuscular injection, 3 doses
  Arms: Group A
Biological: HBV-MPL vaccine (208129)
  Arms: Group C
Biological: Hepatitis B vaccine, experimental formulation — Intramuscular injection, 3 doses
  Arms: Group B

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and reactogenicity of various formulations of recombinant hepatitis B vaccine with different adjuvants in healthy adult volunteers following the 0, 1, 6 months schedule

DETAILED DESCRIPTION:
At the time of conduct of this study, the sponsor GlaxoSmithKline was known by its former name SmithKline Beecham

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 40 years old.
* Written informed consent will have been obtained from the subjects.
* Good physical condition as established by physical examination and history taking at the time of entry.
* Female participants will avoid becoming pregnant during the study period and they will have been on a contraceptive program for at least 2 months before entry

Exclusion Criteria:

* Pregnancy or lactation.
* Serological signs of HBV infection
* Elevated serum liver enzymes
* Any vaccination against hepatitis B in the past.
* Any previous administration of MPL.
* History of significant and persisting hematologic, hepatic, renal, cardiac or respiratory disease.
* Axillary temperature > 37.5°C at the time of injection.
* Any acute disease at the moment of entry.
* Chronic alcohol consumption.
* Any treatment with immunosuppressive or immunostimulant therapy.
* Any chronic drug treatment, which in the investigator's opinion, precludes inclusion into the study.
* History of allergic disease likely to be stimulated by any component of the vaccine.
* Administration of any other vaccine(s) or any immunoglobulin during the study period.
* Simultaneous participation in any other clinical trial.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 1993-06; Primary Completion 1994-07 (Actual); Study Completion 1994-07 (Actual)

PRIMARY OUTCOMES:
Occurrence and intensity of solicited local and general symptoms | 8 days follow-up after vaccination

SECONDARY OUTCOMES:
Anti-HBs antibody concentrations | Months 0, 1, 3, 6, 7, 8 and 12
Occurrence, intensity of unsolicited adverse events | 30-day follow-up after vaccination
Occurrence of serious adverse events | During the study period up to 30 days after last vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Clinical Trials Call Center, Ghent, Belgium